CLINICAL TRIAL: NCT02297360
Title: A 3-Month, Randomized, Double-Blind, Placebo-Controlled Study Evaluating The Ability Of Viviscal Extra-Strength Formulation To Promote Hair Growth And Decrease Shedding In Women With Self-Perceived Thinning Hair
Brief Title: Viviscal Extra-Strength Formulation To Promote Hair Growth And Decrease Shedding In Women With Thinning Hair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ablon Skin Institute Research Center (Other)
Collaborators: Irish Response t/a Lifes2good (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FHOTC 0413
Record Dates: First submitted 2014-11-18; First posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Hair Thinning
Keywords: Hair loss, hair thinning, women, marine protein supplement
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Viviscal Extra-Strength Supplement (Active Comparator): Viviscal Extra-strength tablets. One tablet taken by mouth in the morning and one tablet in the evening with food for 90 days.
  Interventions: Dietary Supplement: Viviscal Extra-Strength Supplement
- Placebo Tablet (Placebo Comparator): Placebo tablets. One tablet taken by mouth in the morning and one tablet in the evening with food for 90 days.
  Interventions: Other: Placebo tablet

INTERVENTIONS:
Dietary Supplement: Viviscal Extra-Strength Supplement — The key ingredient of Viviscal Extra-Strength Supplement is AminoMar C™ marine complex, Equisetum arvense sp. (horsetail), containing a naturally occurring form of silica), Malpighia glabra (acerola cherry) which contains Vitamin C, Biotin and Zinc. The AminoMar C™ is an active ingredient which has been trademarked and comprises of a proprietary blend of shark powder and mollusc powder. It is derived from sustainable marine sources. Viviscal provides essential nutrients to nourish hair naturally from within. The Viviscal supplement is compared to the placebo tablet which contains no active ingredients. One tablet is taken by mouth in the morning and evening with food.
  Arms: Viviscal Extra-Strength Supplement
Other: Placebo tablet — The placebo tablet contains no active ingredients. One tablet is taken by mouth in the morning and evening with food.
  Arms: Placebo Tablet

SUMMARY:
The Viviscal Extra-Strength formulation is an oral food/dietary supplement specifically designed to promote hair growth for women suffering from temporary thinning hair. It does not contain hormones or drugs and has been marketed in Europe for over 15 years. Viviscal Extra-Strength is marketed as Viviscal Maximum Strength in some other territories.

The hypothesis of this clinical research study is that the ingestion of Viviscal Extra-Strength over a three (3) month period will strengthen and promote the growth of terminal hairs in female subjects, ages 21-65 years of age with self-perceived thinning hair associated with poor diet, stress, hormonal influences or abnormal menstrual cycles when compared to using the placebo tablet.

DETAILED DESCRIPTION:
The key ingredient of Viviscal Extra-Strength formulation is AminoMar C™ marine complex, Equisetum arvense sp. (horsetail), containing a naturally occurring form of silica), Malpighia glabra (acerola cherry) which contains Vitamin C, Biotin and Zinc. The AminoMar C™ is an active ingredient which has been trademarked and comprises of a proprietary blend of shark powder and mollusc powder. It is derived from sustainable marine sources. Viviscal provides essential nutrients to nourish hair naturally from within. Viviscal works in many ways over several months of use to improve the appearance of thinning hair.

* Nourishes the hair follicles
* Strengthens and promotes the growth of terminal hairs. Terminal hair is defined as coarse hair, short or long, found on the scalp with minimum cross-sectional diameter of 40 micrometers. Vellus hair is defined as fine, short hairs found on the scalp with maximum cross-sectional diameter of 40 micrometers.
* Supports the growth of hair where it has slowed down or temporarily stopped
* Hair becomes stronger, healthier and more vibrant

Ingestion of Viviscal Extra-Strength over a three (3) month period will strengthen and promote the growth of terminal hairs in female subjects, ages 21-65 years of age with self-perceived thinning hair associated with poor diet, stress, hormonal influences or abnormal menstrual cycles when compared to using the placebo tablet. The primary endpoints will be individual hair counts and favorable analysis using the Nikon CoolPix 4300 with 3GEN Dermlite Foto37 for phototrichogram analysis at the end of the three (3) month period. The secondary endpoints will be statistically significant decreased hair shedding counts with hair washing, favorable improvement in terminal hair diameter measured by the Dino-Lite Digital Microscopic and positive feedback on the Quality of Life and Self-Assessment questionnaires after three (3) months of Viviscal Extra-Strength ingestion.

All patients enrolled must be identifiable throughout the study. The Investigator will maintain a personal list of patient numbers and patient names to enable records to be found at a later date and the list will be stored in a locked cabinet. Subject numbers consist of a 2 digit number from 01 to 60. Patients will be randomized to active or placebo supplements (1:1 ratio) using a randomization table prepared prior to the start of the study by a non-participating staff member at the office of the Investigator. The study blind will not be broken until the end of the study. All test product and placebo will be labeled with subject numbers per the non-participating staff member. Subjects will be assigned a subject number in numerical order as enrolled. Randomization will occur by assignment to either Viviscal Extra-Strength supplement or placebo with 1:1 ratio. Subjects who terminate their study participation for any reason, regardless of whether study medication was used or not, will retain their randomization number.

Visit Procedures Pre-Study Procedures

1. Candidate subjects will be screened with the eligibility requirements by telephone prior to Visit 1.
2. Candidate subjects will be assigned an appointment time for visiting the clinic.

Visit 1: Baseline, Day 0

1. Individuals will be given an informed consent (IC) document & photographic release form, HIPAA form, confidentiality agreement to read. They will have all of their study related questions answered by the Investigator or her designated staff and if they agree, they will sign two copies of the IC/Photography release form, two copies of the HIPAA form, and one copy of the confidentiality agreement. Subjects will be given one copy of the signed IC/Photography release and of the HIPAA agreement to keep, with one copy of each document remaining at the testing facility in the subject's file.
2. Investigator and/or Study Coordinator will review with subject and complete the checklist for all inclusion and exclusion criteria.
3. Investigator and/or Study Coordinator will review with subject and complete the checklist for medical history and concomitant medications.
4. Investigator and/or Study Coordinator will review with subject and complete the General Lifestyle Questionnaire. The General Lifestyle Questionnaire may be found in Appendix V.
5. Subjects will be given a Quality of Life Questionnaire to read and complete. The Quality of Life Questionnaire may be found in Appendix VI.
6. Candidate subjects will receive a brief physical exam, including examination of the scalp, to rule out any immediately observable medical issues and any scalp alopecias/scalp disorders that are unacceptable for qualification. The physical will additionally include vital signs (pulse and blood pressure), weight and height.
7. Candidate subjects of childbearing potential will complete a urine pregnancy test prior to product distribution.
8. Candidate subjects who have completed all the initial paperwork and meet the inclusion/exclusion qualifications (to include findings of the physical exam) will be assigned a unique subject number. Subjects will be randomized to treatment group prior to dispensing the test product.
9. Qualified subjects will have their scalp prepared for digital photography and initial measurements done (see Appendix I).
10. Subjects will have the selected test site photographed (see Appendix I and II).
11. Subjects will have ten (10) terminal hairs in the selected test site cut at the base of the scalp and the diameter of the hairs measured (see Appendix III).
12. Subjects will be instructed to wash their hair at home 24 hours in advance of the study visit. Subjects will have their hair washed (shampooed) with Viviscal Gentle Shampoo over a sink containing cheesecloth (see Appendix IV). The cheesecloth will be positioned to collect shedding hair. The number of hairs collected in the cheesecloth will be counted and recorded. Subjects will be allowed to dry and style their hair.
13. Subjects will be dispensed a three (3) month supply of the test product (three units of Viviscal Extra-Strength or Placebo, as randomized, containing 60 tablets each) and given written and verbal Usage and Lifestyle instructions (see Appendix VIII) and a calendar of future visit. Subjects will be instructed to ingest the test product per Sponsor instructions.

Usage Instructions:

Take two (2) tablets a day, one in the morning and one in the evening; take with water, after food.

Subjects will be instructed to return all empty packets and unused test product at Visit 2.

Lifestyle Instructions:

Subjects will be instructed to maintain their normal hair care routine. Subjects will be instructed to use the same brand/type of hair care products and maintain the same haircut, color and style for the study duration.

Subjects who have color treated hair will also be instructed to have the color treatment performed at the same time interval prior to each visit (ie. If on Visit 1, the color treatment was done one week prior then the color treatment is expected to occur at a similar interval of one week prior to Visit 2).

Subjects will be instructed to come to each visit with clean (shampoo must be done 24 hours prior to the visit) and dry hair.

Subjects will be instructed to use a medically sound form of birth control during the study.

Visit 2: Month 3 (90 days) ± 1 week (7 days)

1. A clinician will ask subjects if they have experienced any changes in their health or taken new/adjusted current medications since the last visit. If an AE or SAE is reported, the examining Investigator will be informed and the appropriate forms will be completed.
2. The test product will be collected and counted for compliance.
3. Subjects will receive a brief physical exam. The physical will include vital signs (pulse and blood pressure).
4. Subjects will complete the Quality of Life Questionnaire and the Self-Assessment Questionnaire (see Appendix VI and VII).
5. Subjects will have their scalp prepared for digital photography (see Appendix I).
6. Subjects will have the selected test site photographed (see Appendix I and II).
7. Subjects will have ten (10) terminal hairs in the selected test site cut at the base of the scalp and the diameter of the hairs measured (see Appendix III).
8. Subjects will be instructed to wash their hair at home 24 hours in advance of the study visit. Subjects will have their hair washed (shampooed) with Viviscal Gentle Shampoo over a sink containing cheesecloth (see Appendix IV). The cheesecloth will be positioned to collect shedding hair. The number of hairs collected in the cheesecloth will be counted and recorded. Subjects will be allowed to dry and style their hair.

All primary and secondary parameters will be collected at Visits 1 and 2. Missing data values will be minimized by intensive training of the interviewers in techniques of clarifying answers and checking questionnaires while participants are on-site. When missing values are identified, several approaches such as rescheduled within 24 hours of completion of tests or interviews will be employed to acquire the necessary data. Missing data will be also examined to assess randomness. Descriptive statistics will be obtained for all variables, tests of normality of continuous measures will be made and data will be examined for homogeneity of variance. An appropriate statistical method will be employed to correct for any abnormalities. All statistical tests will be two-tailed. Differences will be considered statistically significant provided a p-value of 0.05 or less is obtained but other p-values may be evaluated on a case-by-case basis. For each visit, the differences of the two groups from baseline Visit will be tested using analyses of variance with repeated measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Females, ages 21-65 years of age
2. Clinically-determined general good health as determined by responses to the initial study assessment
3. Females with self-perceived thinning hair associated with poor diet, stress, hormone influences or abnormal menstrual cycle as determined on initial study assessment by the Investigator (This will not include patients with medically diagnosed telogen effluvium)
4. Females willing to maintain their normal hair shampooing frequency
5. Females willing to add the provided oral supplement to their current daily routine
6. Females willing to not substantially change their current diet, medications, or exercise routines for the duration of the study. If a subject receives physician guidance during the study to change diet, medications, or exercise routine, the subject will need to notify the clinic as soon as possible
7. Females willing to undergo a brief physical exam to include height, weight, blood pressure, pulse, general physical findings and a scalp exam. The physical exam will occur at Visits 1 and 2
8. Females with Fitzpatrick I-IV photo skin types
9. Willingness to have digital photography of the target area and scalp for hair counts at Visits 1 and 2
10. Willingness to have ten (10) terminal hairs from the target area cut at the base of the scalp for microscopic hair measurements at Visits 1 and 2
11. Willingness to have their hair washed (shampooed) with Viviscal Gentle Shampoo over a sink containing cheesecloth for hair shedding counts at Visits 1 and 2
12. Willingness to maintain a consistent hair cut and hair color throughout the 3 month study period and to come to visits with clean (shampoo must be done 24 hours or more prior to the visit) and dry hair
13. Willingness of subjects who have color treated hair to have the color treatment performed at the same time interval prior to each visit (ie. If on Visit 1 the color treatment was done one week prior then the color treatment is expected to occur at a similar interval of one week prior to Visit 2)

Exclusion Criteria:

1. Females with a known history of intolerance or allergy to fish, seafood/shellfish or acerola
2. Females with any known allergy or sensitivity to any shampoo/conditioner
3. Females who are nursing, pregnant, planning to become pregnant during the study
4. Females with known stressful incident within the last six months (ie. death in family, miscarriage)
5. Females who are participating on any clinical research study at ASIRC or at another research center or doctor's office
6. Females who have recently (within the last 6 months) started the use of hormones for birth control or hormone replacement therapy (HRT). Women currently using hormones for birth control or HRT must have been on a stable dose (6 months or longer) in order to be eligible for the study
7. Females currently using the HairMax light treatment or other light therapy to treat thinning hair
8. Females who have regularly used Rogaine (Minoxidil) within the last 3 months
9. Females who have used prescription drugs known to affect the hair growth cycle within the last 6 months (e.g., hormone-based birth control for less than 6 months, cyproterone acetate, aldactone/spironolactone, Finasteride or any 5-alpha-reductase inhibitor)
10. Females suffering from other hair loss disorders, such as alopecia areata, scarring alopecia, androgenetic alopecia and telogen effluvium as determined on initial study assessment by the Investigator
11. Individuals with self-reported uncontrolled diseases (i.e. diabetes, hypertension, hyperthyroidism, hypothyroidism, etc.). Medical conditions that are under control with or without treatment will be considered on an individual basis by the Investigators
12. Females with self-reported active hepatitis, immune deficiency, HIV or autoimmune disease
13. Females having a known active dermatologic condition which, in the opinion of the examining Investigators, might place the subject at a greater risk or interfere with clinical evaluations (e.g., seborrheic dermatitis, psoriasis, atopic dermatitis, advanced skin cancer, etc.)

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Number of terminal hairs in the target area of the scalp. | 90 days
  The first primary efficacy parameter from the phototrichogram will be the number of terminal hairs in the target area of the scalp. Terminal hair is defined as coarse hair, short or long, found on the scalp with minimum cross-sectional diameter of greater than 40 micrometers. Phototrichogram macrophotographs will be taken of the selected target area of each subject at each visit as specified under the Schedule of Procedures. Digital macrophotography will be performed using a Nikon Coolpix 4300 camera with a 3GEN Dermlite Foto37 system for scalp photography. The macrophotographs are then read by the investigator to determine the terminal hair count.
Number of vellus hairs in the target area of the scalp. | 90 days
  The second primary efficacy parameter from the phototrichogram will be the number of vellus hairs in the target area of the scalp. Vellus hair is defined as fine, short hairs found on the scalp with maximum cross-sectional diameter of 40 micrometers. Phototrichogram macrophotographs will be taken of the selected target area of each subject at each visit as specified under the Schedule of Procedures. Digital macrophotography will be performed using a Nikon Coolpix 4300 camera with a 3GEN Dermlite Foto37 system for scalp photography. The macrophotographs are then read by the investigator to determine the terminal hair count.

SECONDARY OUTCOMES:
Dino-Lite microscopic photographs for terminal hair diameter measurements in the target area | 90 days
  Dino-Lite Microscopic digital photographs to measure the diameter of the hair will be taken of the selected target area of each subject at each visit as specified under the Schedule of Procedures. Ten (10) terminal hairs in the target area will be randomly chosen throughout the area (not all from one direct area) and cut at the surface of the scalp thus not creating any bald patches. The hair diameter will then be measured at 1mm from the cut end of the hair. The ten (10) hair measurements will then be averaged to attain a median hair diameter for the target area.
Hair washing (shampooing) in clinic for hair shedding counts ( | 90 days
  Subjects will be instructed to wash their hair at home 24 hours in advance of study visits 1 and 2. Subjects will then have their hair washed (shampooed) with Viviscal Gentle Shampoo in the office over a sink containing cheesecloth. The cheesecloth will be positioned to collect shedding hair. The number of hairs collected in the cheesecloth will be counted and recorded. Subjects will be allowed to dry and style their hair Subjects will have their hair washed and shedding hairs counted on Visits 1 and 2.
Quality of Life Questionnaire | 90 days
  Questionnaire about the subjects general lifestyle and how their life is affected by thinning hair.
Self-Assessment Questionnaire | 90 days
  Questionnaire is the evaluation of the growth and qualities related to the subjects hair, nails and skin.

CONTACTS AND LOCATIONS:
Overall Officials: Glynis Ablon, MD, FAAD, Principal Investigator — Director Ablon Skin Institute Research Center

REFERENCES:
- [Derived] Ablon G. A 3-month, randomized, double-blind, placebo-controlled study evaluating the ability of an extra-strength marine protein supplement to promote hair growth and decrease shedding in women with self-perceived thinning hair. Dermatol Res Pract. 2015;2015:841570. doi: 10.1155/2015/841570. Epub 2015 Mar 25. PMID 25883641